CLINICAL TRIAL: NCT06469307
Title: Driving Inclusivity, Validity, and Equity in Research Through Strategic Engagement (DIVERSE)
Acronym: DIVERSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Andrew Hantel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-177; K08CA273043 (NIH)
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Blood Cancer; Leukemia
Keywords: Blood Cancer; Leukemia
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DIVERSE Community Advisory Board (CAB) (Other): Enrolled participants will complete:
  * Confidentiality agreement and demographic questionnaire
  * Online training and in-person or remote training with study team
  * Timely DIVERSE review of protocols
  * Audio recorded meeting (in-person, remote, or via phone call) with study team to present review findings
  * Semi-structured exit interview and/or focus group with study staff to provide feedback
  Interventions: Other: DIVERSE Review Process
- DIVERSE Investigators (Other): Enrolled investigator participants will complete:
  * Brief Feedback Survey
  * Request DIVERSE reviews and complete request form
  * Acceptability of Intervention Measure questionnaire
  * Semi-structured exit interview and/or focus group with study staff to provide feedback
  Interventions: Other: DIVERSE Review Process

INTERVENTIONS:
Other: DIVERSE Review Process — A participant and community-based review system for clinical research protocols that elicits and collects feedback on investigator-initiated protocol reviews.
  Other Names: DIVERSE

SUMMARY:
The purpose of this research study is to enhance inclusion and diversity in clinical trial enrollment by training participants to perform and provide feedback through a community-based protocol review process, called DIVERSE.

DETAILED DESCRIPTION:
This research study aims to pilot a protocol review process, called DIVERSE, assessing its feasibility, acceptability, and preliminary efficacy to enhance inclusion and diversity in clinical trial enrollment. Patients and community participants will complete specialized training and provide feedback on clinical trials in development through the DIVERSE process; they will also provide feedback on the process itself. Investigator participants will request review and provide feedback on the DIVERSE process. The study is based on community-based participatory research.

Participation in this research is expected to last about 18 months. It is expected that about 20 patient and community participants and 20 investigators will participate in this research study. The National Cancer Institute and American Society of Clinical Oncology are providing funding for this research study.

ELIGIBILITY:
CAB Participant Inclusion Criteria:

* Age 18 or older
* English speaking
* Ability to understand and willingness to provide oral consent
* DFCI patient who are in remission from a blood cancer >1 year will be preferred.

CAB Participant Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers <18 years old)
* Prisoners.
* Unwilling/unable to agree to maintaining the confidentiality of reviews and clinical trial materials, as outlined in Section 9.1
* Note 1: Patients and non-patient community members who are pregnant are eligible. This is a non-interventional study that meets the definition of minimal risk and poses no greater risk to pregnant individuals or fetuses. Pregnancy status will not be assessed.
* Note 2: English fluency is necessary as protocols being reviewed are written in English and cannot be feasibly translated to other languages within the time period necessary to complete timely reviews.

Investigator Participant Inclusion Criteria:

* Age 18 older
* English Speaking
* Site or Principal investigator
* Not a member of the research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Protocol Review Completion Rate | 18 months
  Feasibility is defined as the proportion of eligible protocols that have completed the DIVERSE review process. The target is a review completion of ≥ 60% of eligible protocols.
Protocol Review Completion Rate Within 35 Days | 18 months
  Feasibility is defined as the proportion of protocols that have completed the DIVERSE review process within 35 days of request. The goal is to have ≥ to 70% of reviews completed within 35 days.
Proportion of Acceptability of Intervention Measure (AIM) Scores of 10 or Greater | 18 months
  Acceptability is defined as the proportion of AIM scores provided by investigators after protocols have been assessed by the DIVERSE review process with ≥ 60% of AIM scores resulting as ≥10 on a scale of 0 - 20, where scores of 10 or above are considered "acceptable" or greater. The AIM is a 4-item, 5-point Likert scale-based measure.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hantel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu